CLINICAL TRIAL: NCT01306097
Title: Evaluating the Impact of 3 Months Daily Zinc Supplementation on Incidence of Severe and Recurrent Diarrhea in 6 to 36 Months Age Children
Brief Title: Zinc Supplementation and Severe and Recurrent Diarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Marzie Barchinejad, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Zinc supplementation
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2009-01

CONDITIONS: Diarrhea
Keywords: Zinc Supplement; Diarrhea; Sever Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Zinc Sulfate; Zinc

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zinc sulfate (Experimental): daily zinc supplementation for 3 months. (10mg daily for under 1 years old children and 20mg daily for above 1 years old children)
  Interventions: Drug: Zinc Supplement

INTERVENTIONS:
Drug: Zinc Supplement — 10mg daily for under 1 years old children and 20mg daily for above 1 years old children
  Other Names: Zinc sulfate; Oral Zinc

SUMMARY:
Evaluating the impact of 3 months daily zinc supplementation on incidence of severe and recurrent diarrhea in 6 to 36 months age children in Bandarabbaas

DETAILED DESCRIPTION:
Evaluating the impact of 3 months daily zinc supplementation on incidence of severe and recurrent diarrhea in 6 to 36 months age children in Bandarabbaas in 2009

ELIGIBILITY:
Inclusion Criteria:

* All 6 to 36 months old children without diarrhea at the time of study and without disease such as celiac
* Inflammatory bowl disease and hypersensitivity to milk

Exclusion Criteria:

* Diarrhea at the time of the study and background disease such as celiac, IBD or hypersensitivity to milk

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Diarrhea | 1 years
  Incidence, Duration and frequency

SECONDARY OUTCOMES:
Admission for diarrhea | 1 year
  Total number of admissions during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Marzie Barchinejad, Principal Investigator — Hormozgan University of Medical Sciences
Locations (1):
- Hormozgan University of medical sciences, Bandar Abbas, Hormozgan, Iran

REFERENCES:
- [Derived] Imdad A, Rogner J, Sherwani RN, Sidhu J, Regan A, Haykal MR, Tsistinas O, Smith A, Chan XHS, Mayo-Wilson E, Bhutta ZA. Zinc supplementation for preventing mortality, morbidity, and growth failure in children aged 6 months to 12 years. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD009384. doi: 10.1002/14651858.CD009384.pub3. PMID 36994923